CLINICAL TRIAL: NCT06946082
Title: It is to Examine the Relationship Between Upper Extremity Motor Function, Trunk Control, Motor Imagery.
Brief Title: The Effect of Upper Extremity Motor Function, Trunk Control and Motor Imagery Ability on Turkish Language Skills in Individuals With Stroke
Status: Recruiting | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Emine Timur, Researcher/Student, Izmir Bakircay University
Other Study IDs: bakircay-timur
Record Dates: First submitted 2025-04-15; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hemiplegia; Aphasia; Stroke; Trunk; Upper Limbs; Motor Imagery
MeSH Terms: conditions — Hemiplegia; Aphasia; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A large number of people have a stroke each year and it is a major cause of disability worldwide. Upper limb motor impairments, aphasia, body control problems and decreased motor imagery ability are common after stroke. Although there are studies showing that these impairments may be related to each other, there is no comprehensive study examining the relationship between Turkish language skills and these motor functions. The aim of this study was to evaluate the relationship between Turkish language skills and upper extremity motor function, trunk control and motor imagery ability in stroke patients.

DETAILED DESCRIPTION:
Each year, approximately 800,000 individuals experience a new or recurrent stroke. Although mortality rates have declined in recent years, the number of stroke survivors has increased, making stroke the third most common cause of disability worldwide.

In stroke patients, both upper extremity (UE) motor impairment and language function disorders are frequently observed. These two types of post-stroke dysfunctions are among the most prominent neuropsychological deficits: UE motor impairment occurs in approximately 80% of stroke patients, aphasia in 21-38%, and both conditions co-occur in about 24% of cases. Upper extremity motor impairment combined with aphasia affects social participation and quality of life and is also associated with many comorbidities, potentially leading to a poor prognosis. Due to their anatomical proximity, ischemia or hemorrhage in the middle cerebral artery (MCA) often results in UE motor impairments and non-fluent aphasia. Hybbinette et al. confirmed through a small sample study that apraxia of speech and aphasia commonly co-occur with hand motor deficits in patients with left hemisphere stroke.

Aphasia is defined as acquired neurological damage to areas of the brain responsible for understanding and producing language and symbols. This damage disrupts the connection between speaking, thinking, and interpreting. A recent prospective study by Grönberg and colleagues revealed that despite a decrease in ischemic stroke rates over the last decade, 30% of patients with acute ischemic stroke still experience aphasia.

Post-stroke aphasia is a major disability that negatively impacts rehabilitation and overall stroke outcomes. It is one of the most detrimental conditions affecting health-related quality of life, associated with high risk of depression and reduced likelihood of returning to work. Accurate knowledge of the symptoms and factors associated with aphasia is essential for optimal care.

One of the most common issues in stroke patients is upper extremity motor dysfunction. One-third of stroke survivors continue to experience deficits even six months post-stroke. Another disabling consequence of stroke is impairment in trunk motor control and balance. One of the main roles of the trunk is to support limb movements by activating before or during goal-directed actions. However, in stroke patients, motor impairment leads to decreased or delayed trunk muscle activation, which causes deviations in limb movements and postural abnormalities. These abnormal movement patterns and posture, resulting from stroke, are the primary cause of early trunk control disorders. Trunk dysfunction also affects respiration and, consequently, phonation, which is known to impact speech abilities in stroke patients. This suggests that trunk control plays an important role in predicting the efficiency of post-stroke rehabilitation and functional recovery.

Imagery refers to mentally creating or recreating an experience or knowledge. Motor imagery (MI) is the process of mentally simulating a movement without physically performing it. During imagery, the neuronal activity that occurs between the cerebral cortex, cerebellum, and brainstem is similar to that during actual movement.

One major challenge in using motor imagery is determining the extent to which a person can form mental representations of movement. After stroke, this becomes more problematic. The slowing down of imagery after stroke suggests that the temporal characteristics of imagery may be altered. These findings indicate that some patients may not be able to use motor imagery at all. Therefore, evaluating imagery ability in stroke patients is crucial.

One study comparing stroke survivors and a control group found that stroke patients experienced difficulties in understanding and performing tasks related to motor imagery.

Cayol et al. (2020) aimed to investigate the relationship between performance on a motor imagery task and word-definition task in adolescents. The results indicated that MI ability predicts language processing skills. This finding aligns with literature suggesting the role of MI in representing action-related concepts in the brain. The correlation between MI ability and language processing skills implies that the brain can represent action-related information more effectively.

Additionally, Taub and colleagues observed that stroke patients often fail in upper extremity motor function tasks, leading them to avoid using the affected limb-a phenomenon known as "learned non-use." In such cases, both the willingness to move and the memory of movement imagery for the affected limb may be impaired. Patients make repeated errors, which reduces motivation to use the limb, hindering recovery of motor function.

The collected evidence indicates that language skills, upper extremity motor function, trunk control, and motor imagery ability are all affected in stroke patients. Several studies suggest potential relationships between these domains. However, no comprehensive research has been conducted examining the relationship between these three domains and language skills in Turkish.

This study aims to contribute to multidisciplinary rehabilitation approaches by offering new perspectives and supporting the development of combined evaluation and treatment methods in the future.

Although there are studies in various languages examining the relationship between upper extremity motor function and language ability in stroke patients, there is a lack of research involving Turkish-speaking individuals. Exploring how these two areas interact specifically in Turkish speakers may provide important insights for recovery.

Furthermore, no studies have examined the impact of language skills on trunk control and motor imagery ability. To fill this gap, our study aims to evaluate the relationship between Turkish language skills and upper extremity motor function, trunk control, and motor imagery in stroke patients. Understanding this connection will be a valuable guide in rehabilitation processes.

Therefore, our goal is to assess the impact of upper extremity motor function, trunk control, and motor imagery ability on Turkish language skills in individuals who have experienced a stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Stroke onset more than 1 week
* Not having practiced imagery before
* Being a native speaker of Turkish
* Standardized Mini Mental Test (SMMT) Score of 24 and above
* History of cerebrovascular events
* Not having any neurological disorder other than stroke
* The ability to grasp and hold a 2.5 cm cube

Exclusion Criteria:

* No consent from the family or person
* Having had a stroke before
* Severe hearing or vision loss
* Individuals are excluded if they have other primary medical conditions that may affect language and motor functions (e.g. brain tumor, Parkinson's disease, severe post-stroke depression, Alzheimer's disease) or have undergone surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted with individuals who have had a stroke and are 18 years of age or older. Participants will be individuals who have had a stroke at least 1 week ago, who have not received motor imagery practice before, whose native language is Turkish, and whose cognitive competence has been confirmed by the Standardized Mini Mental Test (SMMT) (≥24 points). In addition, only individuals with a history of cerebrovascular events will be included.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Aphasia Language Assessment Test (ADD) | Baseline (upon enrollment)
  The Aphasia Language Assessment Test was developed by Maviş and Toğram. It is a language test that allows diagnosing aphasia, determining the type of aphasia, determining the performance of the individual with aphasia in all language areas and selecting appropriate therapy goals for the individual. The Aphasia Language Assessment Test consists of 8 subtests assessing speech fluency, auditory comprehension, repetition, naming, reading, speech acts, grammar and writing. Correct and independent responses are scored as 2; incomplete, inadequate or assisted responses as 1 and incorrect responses or no response as 0.
GAT-2 (Gulhane Aphasia Test) | Baseline (upon enrollment)
  This test consists of six parts and assesses the individual's awareness, comprehension (speech comprehension, reading comprehension), oral-motor skills, automatic speech, repetition and naming skills. This test also determines whether the individual diagnosed with aphasia is accompanied by dysarthria, apraxia or paraphasia in language production. Hearing comprehension is evaluated with 20 items, reading comprehension with 15 items, repetition with 6 items and naming with 13 items. The score of each section is expressed as a percentage. The total aphasia score is obtained by summing the scores of all sections (minimum 0, maximum 600 points). A lower aphasia score indicates more severe aphasia. A score of 40% or less on at least three sections indicates moderate-to-severe aphasia. However, the GAT only gives a numerical value for aphasia, and aphasia cannot be typed.

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment Scale (FMA-UE) | Baseline
  The Fugl Meyer Upper Extremity Assessment Scale is a performance-based scale (Van Wijck FM et al 2001, Gladstone D et al 2002). The test consists of reflex activity, flexor and extensor synergy, combined synergistic movements, non-synergistic movements, normal reflex activity, wrist and hand assessment, coordination and speed assessment. It consists of 33 items in total and each item is scored between 0 and 2 points (0: unable, 1: partially able, 2: fully able). The total score is 66.
Upper Extremity Activity Test | Baseline
  The upper extremity activity test is a 19-item performance test used to evaluate upper extremity function in stroke survivors and patients after brain injury. It was developed by Lyle in 1981. The test is divided into four subscales: coarse grasp, fine grasp, fingertip grip and gross movement. It is organized hierarchically from the most difficult task to the least difficult task. It is suggested that normal movement in the most difficult task will be an indicator of successful performance in the following tasks and will increase the efficiency of the test. Task performance is assessed on a 4-point scale ranging from 0 (no movement) to 3 (movement is performed normally). In the ARAT, scores range from 0-57 and a high score indicates no dysfunction in the upper limb.
Body Disorder Scale | Baseline
  It is a test developed to evaluate the trunk control of stroke patients. It includes 3 subheadings evaluating static sitting balance, dynamic sitting balance and coordination. Static sitting balance includes 3 questions, dynamic sitting balance includes 10 questions and coordination includes 4 questions. It is scored between 0 and 23. 0 is the lowest value and 23 is the highest value and indicates good trunk control. It is important in terms of evaluating the quality of trunk movements, examining the development and shaping the treatment. This test, which has proven its validity and reliability in our country as in many countries, provides a detailed examination of trunk control, which is a very important part of postural control and balance.
Functional Independence Scale (FIM) | Baseline
  The Turkish version of the Functional Independence Scale (FIM) was used to assess functional independence in activities of daily living. The FIM analyzes two different aspects of disability, motor and cognitive functions. It consists of six functional sections: self-care, sphincter control, mobility, locomotion, communication and social perception. In the FIM, a total of 18 activities are assessed for functional independence using a seven-point scale for each. Each item is scored from 1-7 points in proportion to the amount of assistance received (1 point: fully assisted, 7 points: fully independent). The minimum score is 18 and the maximum score is 126.
Movement Imagery Survey-3 (MIS) | Baseline
  The Movement Imagery Questionnaire-3 is the most up-to-date version of the Movement Imagery Questionnaire and the Movement Imagery Questionnaire - Revised, 2nd Edition. The 12-item questionnaire assesses external, internal and kinesthetic imagery separately. The questionnaire will be used in this study to directly assess motor imagery. During the administration of the questionnaire, individuals will be asked to first physically perform 4 different movements and then to visualize once with external imagery, once with internal imagery and once with kinesthetic imagery. It is scored on a scale from 1 to 7. A score of 1 means "very difficult to see/feel", while a score of 7 means "very easy to see/feel"
Kinesthetic and Visual Imagery Questionnaire-20 (KGIA-20) | Baseline
  It is a valid and reliable tool used to assess imagery ability. The KGIA-20 questionnaire has visual and kinesthetic sections. This questionnaire allows clinicians and physiotherapists to quickly assess imagery in a sitting position. A trained and experienced practitioner is needed to administer the questionnaire. The questionnaire includes a total of 20 topics, 10 visual and 10 kinesthetic. With the questionnaire, the intensity level of imagery is recorded on a 5-point Likert scale (5= a vivid image appears; 1= no image or sensation appears). A high score is accepted as an indicator of good imagery level (21) The highest score that can be obtained separately for kinesthetic imagery and visual imagery is 85 and the lowest score is 17. At the end of the questionnaire, the sum of the kinesthetic imagery and visual imagery scores is obtained and the highest score is 170 points and the lowest score is 34 points. Higher scores on the KGIA indicate better motor imagery ability.
Box and Block Test: | Baseline
  The Box and Block Test is a test developed to measure gross manual skill. In this study, unlike the classical method, the time taken to collect 15 blocks will be recorded instead of the number of blocks collected in a limited time. The aim is to assess mental chronometry ability rather than manual skill. The test starts from the position where the blocks are on the affected side of the individual. First, 15 blocks are physically moved and the time is recorded (MET). Then, the materials are removed and the same task is performed with mental imagery and the time is again recorded (MIT). Mental chronometry ability is calculated by the formula (MET-MIT)/MET; a result closer to 0 indicates better performance.
Hand Lateralization Test | Baseline
  In the Hand Lateralization Test, individuals will be shown visuals of the right and left hand from 4 surfaces and 12 angles and asked about the direction of the hand. The test is performed in a sitting position with the hands in the lap. The sum of true-false, right, left, affected and unaffected side correct numbers will be recorded. Evaluation will be done with the mobile application called 'Orientate'.
Standardized Mini Mental Test | Baseline
  The Standardized Mini-Mental Test is a widely used test of cognitive function and consists of 11 items grouped under 5 main headings: orientation, memory, attention and calculation, recall, and language. It is evaluated on a total of 30 points. Scores between 24-30 points will be considered normal, 18-23 points will be considered mild dementia, and scores of 17 and below will be considered severe dementia, and individuals with an SMMT score of 24 and above will be included in our study.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)